CLINICAL TRIAL: NCT05583188
Title: Neoadjuvant Soft Tissue Ablation Utilizing Aliya™ Pulsed Electric Fields With Systemic Therapy in Early-Stage Resectable Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Neoadjuvant Aliya™ PEF Soft Tissue Ablation With Systemic Therapy in Early-Stage Resectable NSCLC
Acronym: VIGOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategic
Sponsor: Galvanize Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-00012
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: NSCLC
Keywords: Lung Neoplasms; Thoracic Neoplasms; Lung Diseases; Antineoplastic Agents; Immunologic Factors; Immune Checkpoint Inhibitors; Nivolumab; Gemcitabine; Cisplatin; Docitaxel; Pemetrexed
MeSH Terms: conditions — Lung Neoplasms; Thoracic Neoplasms; Lung Diseases | interventions — Nivolumab; Carboplatin; Pemetrexed; Gemcitabine; Paclitaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Aliya PEF ablation (Experimental): Pulsed electric field treatment using the Aliya System
  Interventions: Device: Aliya Pulsed Electric Fields (PEF) ablation; Drug: Nivolumab plus Platinum Doublet Chemotherapy; Drug: Standard of care neoadjuvant therapy; Other: Surgical Resection

INTERVENTIONS:
Device: Aliya Pulsed Electric Fields (PEF) ablation — Patients will undergo PEF ablation
Drug: Nivolumab plus Platinum Doublet Chemotherapy — If EGFR/ALK mutation negative, patients will receive standard of care dosing of three cycles of nivolumab at a dose of 360 mg every three weeks along with a platinum-based chemotherapy doublet (cisplatin or carboplatin plus pemetrexed for adenocarcinoma, cisplatin or carboplatin plus docetaxel, paclitaxel, or gemcitabine for squamous NSCLC) post-PEF ablation followed by resection.
  Other Names: Carboplatinum; Cipsplatin; Pemetrexed; Gemcitabine; Paclitaxel
Drug: Standard of care neoadjuvant therapy — Patients not eligible for neoadjuvant nivolumab plus chemotherapy will receive standard of care systemic therapy post-PEF ablation followed by resection.
  Other Names: Carboplatinum; Cipsplatin; Pemetrexed; Gemcitabine; Paclitaxel; Vinorelbine
Other: Surgical Resection — Patients not eligible for systemic therapy will receive definitive surgery without neoadjuvant therapy as per institutional standard of care post-PEF ablation.

SUMMARY:
A prospective, single-arm, non-randomized, multi-center, open-label study following patients with resectable stage IIB to IIIA non-small cell lung cancer after Pulsed Electric Fields (PEF) ablation who may be candidates for standard of care neoadjuvant use of checkpoint inhibitor (nivolumab) treatment plus platinum doublet chemotherapy.

DETAILED DESCRIPTION:
This study is designed to evaluate the pathologic response of soft tissue ablated with Pulsed Electric Fields (PEF) in patients with resectable stage IIB to IIIA NSCLC who may be candidates for standard of care neoadjuvant use of checkpoint inhibitor (nivolumab) treatment plus platinum doublet chemotherapy. The study will enroll adult patients with suspected or confirmed 8th ed. Stage IIb-IIIA non-small cell lung cancer (NSCLC) who are surgical candidates and have not yet received treatment for NSCLC. PEF ablation may be performed in conjunction with the clinically appropriate approach to collect standard of care biopsy samples to confirm disease progression. PEF ablation will be delivered via percutaneous approach utilizing the Galvanize Aliya™ System and the percutaneous Aliya Ablation Device.

SOC neoadjuvant systemic treatment will be delivered following PEF ablation delivery according to EGFR and ALK mutation status, tumor histology, and surgical candidacy. Patients will undergo surgical resection per standard of care.

The study will consent up to 15 adult patients in order to accrue at least five (5) patients who have completed surgical resection after receiving neoadjuvant therapy with nivolumab plus chemotherapy following PEF ablation.

The remaining patients (up to 10) not eligible for neoadjuvant nivolumab plus chemotherapy will receive either SOC systemic therapy post-PEF ablation followed by resection or, if not eligible for systemic therapy, will receive definitive surgery without neoadjuvant therapy as per institutional SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older
2. Radiographic findings consistent with a lesion with high pre-procedure probability of malignancy as determined by the investigator to be NSCLC 8th Ed. stage IIB- IIIA cancer or biopsy-confirmed NSCLC 8th Ed. stage IIB-IIIA and lesion size ≤ 5 cm in greatest dimension
3. Lesion is targetable for biopsy and PEF delivery per investigator opinion
4. Patient deemed able to complete neoadjuvant therapy according to their EGFR/ALK mutation status and specific histology (if clinically appropriate) and per the manufacturer's systemic therapy labeling
5. Patient has been deemed a potential candidate for definitive lung tissue resection by a qualified study investigator
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
7. Patient is able to adhere to protocol requirements
8. Patient is able to tolerate general anesthesia
9. Patient is cleared to undergo paralytic anesthesia
10. Patient has provided informed consent

Exclusion Criteria:

1. Presence of advanced, inoperable, or metastatic disease
2. Radiographically suspicious findings for stage IIIA patients indicating a single mediastinal lymph node > 3 cm or multiple mediastinal lymph nodes and, therefore, potentially inoperable
3. Patient has recurrent NSCLC or has previously been treated for NSCLC
4. Patient has received chemotherapy or any other cancer therapy in 2 years prior to PEF ablation
5. Prior treatment with any drug that targets T cell co-regulatory pathways (such as checkpoint inhibitors) in 2 years prior to PEF ablation
6. Patient requires or is likely to require a pneumonectomy
7. Patient has received any vaccine against infectious diseases (e.g., influenza, COVID-19, varicella, etc.) within 30 days of PEF procedure Patient is unable or unwilling to complete all required screening and/or follow-up assessments
8. Patient is currently enrolled in another interventional clinical trial or is receiving treatment with an investigational medication or medical device that conflicts with the study protocol

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Pathologic response | Surgical resection
  Pathologic response (percentage of residual viable tumor cells) of the resected lesion ablated with PEF and in resected lymph nodes in patients who received standard of care neoadjuvant nivolumab plus chemotherapy prior to resection.

SECONDARY OUTCOMES:
Rate of R0 resection | Surgical resection
  R0 - no cancer cells seen microscopically at the primary tumor site

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, MD, Study Chair — Chief Medical Officer
Locations (3):
- United States (3):
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plan of data sharing

REFERENCES:
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Background] Hellmann MD, Chaft JE, William WN Jr, Rusch V, Pisters KM, Kalhor N, Pataer A, Travis WD, Swisher SG, Kris MG; University of Texas MD Anderson Lung Cancer Collaborative Group. Pathological response after neoadjuvant chemotherapy in resectable non-small-cell lung cancers: proposal for the use of major pathological response as a surrogate endpoint. Lancet Oncol. 2014 Jan;15(1):e42-50. doi: 10.1016/S1470-2045(13)70334-6. PMID 24384493
- See also: CheckMate 816 Clinical Study — https://clinicaltrials.gov/ct2/show/NCT02998528